CLINICAL TRIAL: NCT02478697
Title: Tobacco Treatment for Employable Californians (TTEC), Improving Employability Partnership: Alliance to Curb Tobacco (Total IMPACT)
Brief Title: Tobacco Treatment for Employable Californians, Total IMPACT Study
Acronym: TTEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: San Francisco Employment Development Department (Unknown); CareerPoint Marin (Other); JobTrain (Unknown); Marin City Community Development Corporation (Unknown); Oakland Employment Development Department (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24RT-0035
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Tobacco Dependence
Keywords: tobacco smoking behavior; employment; job-seeking; tobacco cessation; transtheoretical model; behavior change
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tobacco Treatment (Experimental): The tobacco treatment includes: (a) the ProChange ExpertSystem, a Transtheoretical-model (TTM) tailored, computer-assisted web-delivered program focused on increasing intrinsic motivation, (b) a stage-tailored treatment manual with goal setting for quitting tobacco, and (c) education on proper use of nicotine replacement therapy (NRT, patch plus gum or lozenge) with guidance on obtaining low-cost or free NRT through MediCal, private insurance plans, and community programs.
  Interventions: Behavioral: ProChange ExpertSystem
- Usual Care (No Intervention): Usual care includes: completing the study assessments at baseline, 3- and 6-months and receiving referrals to tobacco treatment in the community, including the state quitline, in line with the public health "Ask, Advise, Refer" model of tobacco cessation intervention.

INTERVENTIONS:
Behavioral: ProChange ExpertSystem — The computer program assesses stage of change and TTM constructs of temptations, decisional balance, and processes of change. Repeat intervention contacts occur at baseline, 3- and 6-months follow-up, providing iterative computerized feedback reflecting prior responses with encouragement for quitting smoking and relapse prevention.
  Other Names: ProChange
  Arms: Tobacco Treatment

SUMMARY:
Previous findings indicate elevated risk for tobacco use among adults in California who are unemployed and seeking work. In a pilot study, tobacco use was associated with a longer duration of time out of work. This community-based participatory research study aims to deliver and evaluate the impact of a web-based job seeker tailored tobacco cessation intervention vs. a control group in the San Francisco Bay Area. This research investigates whether an employment-centered tobacco treatment intervention is efficacious in supporting abstinence and also associated with more timely engagement of employment.

DETAILED DESCRIPTION:
PLEASE NOTE: The grant for this project was approved under the title "Tobacco Treatment for Employable Californians," abbreviated "TTEC."

However, as this study is being run under the principles of community- based participatory research, the Stanford team provided the community advisors and representatives of the recruitment sites the opportunity to create a name they felt better conveyed the interests and goals of the study to potential participants. As such, the term Total IMPACT Study is used on all participant-facing materials.

Dr. Prochaska will oversee study procedures for participant recruitment, informed consent, data collection, analysis, and dissemination. IRB approved study flyers and e-communications will promote the study with a central study contact phone number and email address held by the study coordinator. The study will follow the Dillman method for electronic communications inviting and encouraging potential respondents to participate. For systematic data collection and storage, all assessments will be conducted using Qualtrics or RedCap for online data collection with data encryption for added security protection.

Face-to-face informed consenting procedures occur onsite at the employment agencies. Some participants may call in and get preliminarily screened for eligibility over the phone, but will be directed to meet with on-site staff to begin the consent process. Hired and trained field research study staff will be recent job-seeking clients from the agencies who will complete the informed consenting procedures with participants, obtain collateral contact information for follow-up contacts, and provide participants with a study ID code and the website URL for completing the online survey. The collateral contact information will be used if research staff cannot reach the participant directly. Study staff may ask collateral contacts for updated contact information as well as updated smoking and/or employment status (e.g., "Has [name] been smoking recently?" "Do you know if [name] is currently working?)

Study eligibility will be defined as unemployed and job seeking at a participating America's Job Centers of California (AJCC) organization and currently smoking 1 or more cigarettes daily and at least 100+ cigarettes in one's lifetime with a carbon monoxide (CO) breath sample of 10 ppm or greater. The CO sample will be taken prior to consenting potential participants. Participants must be 18 years or older, English literate, able to provide at least three collateral sources of contact for follow-up assessments, and not immediately planning to relocate out of California (though researchers would continue to follow-up with participants who move out of area, and the research team has demonstrated success with doing so in prior studies). Dual use of e-cigarettes will not be an exclusion criterion.

If a participant meets all eligibility criteria, the baseline assessment will be completed on-site at the employment agency.

A computer-generated stratified random assignment program will randomize individuals based on their recruitment location, heaviness of smoking (> 1 pack/week), and stage of change, the last two variables known to be related to outcomes and addressed by the intervention. Participants will be given study materials appropriate to their assigned study condition directly after completing the baseline survey on-site.

The online surveys will not collect any personal identifying information. Assessments will be conducted at baseline and 3- and 6-months follow-up. The surveys will take about 40 minutes to complete. If participants cannot come in person to do the survey, research staff will send them the URL link, complete it over the phone, or send a modified version in the mail.

As part of data collection, participants will be asked to provide a resume or curriculum vitae at the baseline interview, either as a hard copy or by email, which will be de-identified (participant name and address removed). The resumes will not be shared with staff of the employment service facilities. In a more detailed manner than captured by the self-report online survey, the resumes will provide useful information on prior employment (# of jobs, industry, positions held, length of employment) and education as well as an indication of participant communication/organization skills in self-presentation of employment strengths. Participants will have the option to opt out of providing the resume.

The two study conditions are: Tobacco Intervention (n=180) and Usual Care Control group (n=180).

The tobacco treatment includes: (a) a Transtheoretical-model (TTM) tailored, computer-assisted web-delivered program focused on increasing intrinsic motivation, (b) a stage-tailored treatment manual with goal setting for quitting tobacco, and (c) education on proper use of nicotine replacement therapy (NRT, patch plus gum or lozenge) with guidance on obtaining low-cost or free NRT through MediCal, private insurance plans, and community programs.

The computer program assesses stage of change and TTM constructs of temptations, decisional balance, and processes of change. Repeat intervention contacts occur at baseline, 3- and 6-months follow-up, providing iterative computerized feedback reflecting prior responses with encouragement for quitting smoking and relapse prevention.

Usual care: Participants complete the study assessments at baseline, 3- and 6-months and will receive referrals to tobacco treatment in the community, including the state quitline, in line with the public health "Ask, Advise, Refer" model of tobacco cessation intervention.

Measures:

Primary Tobacco Outcome: At baseline and follow-ups, past 7-day use of conventional cigarettes, alternative tobacco (smokeless, snus), and electronic nicotine devices (ENDS, e.g., e-cigarettes) with details on cigarettes/day, frequency, brand, flavor, strength, and quit attempts are assessed. For biochemical verification, participants reporting 7-day PPA at follow-up will have an expired CO sample evaluated using a Bedfont Smokerlyzer. Participants with CO < 8 ppm indicating nonsmoking will provide a saliva sample for testing with of cotinine with an Accutest® NicAlertTM test strip at the 3- and 6-month follow-ups. Salivary cotinine levels < 15 ng/ml will confirm nonsmoking. Additionally, participants reporting being quit will be asked to provide a urine sample to test for the presence of anabasine (if they have quit smoking but are still using nicotine replacement or another nicotine containing product). Anabasine is an alternative indicator of tobacco exposure that is separate from nicotine.

For participants lost to follow-up or unable to return for biochemical verification, a saliva cotinine test will be mailed, along with a prepaid envelope to return their results to study staff in.

Secondary Tobacco Outcomes: 3-mo prolonged abstinence from the 3- to 6-mo assessment, applying NHLBI's definition of relapse (i.e., smoking on 7 consecutive days or smoking at least once each week over 2 consecutive weeks);42 reduction in cigarettes per week; and given the uncertainty in the field with respect to how to treat ENDS, will examine the proportion of the sample abstinent from conventional cigarettes and all tobacco, allowing for ENDS use.

The observational Personal Professional Presence (P3) checklist scale is currently being pilot tested, and evaluation in relation to measured CO levels will be analyzed as an indicator of treatment compliance and used as an instrumental variable in tobacco outcome analyses.

Employment Outcomes: The primary employment outcome of interest is how quickly participants find employment, measured in weeks. Time out of work is assessed at baseline.

Secondary employment outcomes of interest are: employment status at each follow-up and employment secured at any point in time during the study assessed at 3- and 6-month follow-up. Additional details are obtained on type of position, pay/salary, fit between the secured and desired position, and changes in employment over time. The number of on-phone and in-person interviews also are recorded.

Descriptive Measures. To describe the sample researchers will measure participant gender; age; ethnicity/race; education (years); income; subjective social standing in one's self-defined community and in the broader US; stability of housing; height/weight (BMI); employment history, including days since last regular employment; job search strategies; criminal history; home smoking rules; exposure to secondhand smoke; years of smoking; Fagerström Test for Nicotine Dependence; Stage of Change categorized as precontemplation, contemplation, preparation, action, and maintenance; and Thoughts about Abstinence assessing desire, expectancy of success, anticipated difficulty, and abstinence goal. Assessments of co-occurring substance use and abuse include ASI items 30 day substance use, AUDIT, and DAST. The staging health risk assessment assesses additional health risks and future behavioral targets.

Lastly, a social network stem question where participants are asked to identify up to 10 individuals (alters) in their social network who currently support them in their job search, indicating the strength of the connection, the frequency of contact, and the individuals' job and smoking status. Additional questions about the type of employment (field of employment and position within company) each alter has will be included.

Process Measures. At baseline and each follow-up use of in-study and out-of-study cessation methods including dose, duration, and formulation of NRT, varenicline, bupropion, written materials, provider advice and counseling, quitlines, and other community cessation programs will be assessed. Assessment of study treatment acceptability will be completed by participants in both conditions with 5-items tapping relevance, usefulness, feasibility, level of engagement, perceived fit measured on 5-point Likert scales.

ELIGIBILITY:
Inclusion Criteria: Study eligibility will be defined as unemployed and job seeking at a participating America's Job Centers of California (AJCC) organization and currently smoking 1 or more cigarettes daily and at least 100+ cigarettes in one's lifetime with a carbon monoxide (CO) breath sample of 10 ppm or greater. The CO sample will be taken prior to consenting potential participants. Participants must be 18 years or older, English literate, able to provide at least three collateral sources of contact for follow-up assessments, and not immediately planning to relocate out of California (though researchers would continue to follow-up with participants who move out of area, and have demonstrated success with doing so in prior studies). Dual use of e-cigarettes will not be an exclusion criterion.

Exclusion Criteria: Failure to meet inclusion criteria; non-job-seeking, persons employed or underemployed, occasional/non-daily smokers, daily smokers with carbon monoxide readings less than 10ppm, nonsmokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Smoking Status: 7-day point prevalence abstinence | 3-months follow-up
  Past 7-day use of conventional cigarettes, alternative tobacco (smokeless, snus), and electronic nicotine devices (ENDS, e.g., e-cigarettes) with details on cigarettes/day, frequency, brand, flavor, strength, and quit attempts. For biochemical verification, participants reporting 7-day PPA at follow-up will have an expired CO sample evaluated using a Bedfont Smokerlyzer. Participants with CO < 8 ppm indicating nonsmoking will provide a saliva sample for testing with of cotinine with an Accutest NicAlertTM test strip. Salivary cotinine levels < 15 ng/ml will confirm nonsmoking. Additionally, participants reporting being quit will be asked to provide a urine sample to test for the presence of anabasine (if they have quit smoking but are still using nicotine replacement or another nicotine containing product).
Smoking Status: 7-day point prevalence abstinence | 6-months follow-up
  Past 7-day use of conventional cigarettes, alternative tobacco (smokeless, snus), and electronic nicotine devices (ENDS, e.g., e-cigarettes) with details on cigarettes/day, frequency, brand, flavor, strength, and quit attempts. For biochemical verification, participants reporting 7-day PPA at follow-up will have an expired CO sample evaluated using a Bedfont Smokerlyzer. Participants with CO < 8 ppm indicating nonsmoking will provide a saliva sample for testing with of cotinine with an Accutest? NicAlertTM test strip. Salivary cotinine levels < 15 ng/ml will confirm nonsmoking. Additionally, participants reporting being quit will be asked to provide a urine sample to test for the presence of anabasine (if they have quit smoking but are still using nicotine replacement or another nicotine containing product).
Time to find employment (weeks) | 6-months
  How quickly participants find employment, measured in weeks

SECONDARY OUTCOMES:
3-month Prolonged Abstinence | 6-months follow-up
  3-mo prolonged abstinence from the 3- to 6-mo assessment, applying NHLBI's definition of relapse (i.e., smoking on 7 consecutive days or smoking at least once each week over 2 consecutive weeks);42 reduction in cigarettes per week; and given the uncertainty in the field with respect to how to treat ENDS, will examine the proportion of the sample abstinent from conventional cigarettes and all tobacco, allowing for ENDS use.
Employment Status | 3-months follow-up
  Whether a participant is working or not at the time of assessment.
Employment Status - Current | 6-months follow-up
  Whether a participant is working or not at the time of assessment.
Employment Status - Within study period | 6-months follow-up
  Whether the participant was able to secure employment at any point within the study.

CONTACTS AND LOCATIONS:
Overall Officials: Judith J Prochaska, PhD, MPH, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - JobTrain, Menlo Park, California
  - San Francisco Employment Development Department, San Francisco, California
  - Marin Employment Connection, San Rafael, California

REFERENCES:
- [Background] Hall SM, Tsoh JY, Prochaska JJ, Eisendrath S, Rossi JS, Redding CA, Rosen AB, Meisner M, Humfleet GL, Gorecki JA. Treatment for cigarette smoking among depressed mental health outpatients: a randomized clinical trial. Am J Public Health. 2006 Oct;96(10):1808-14. doi: 10.2105/AJPH.2005.080382. PMID 17008577
- [Background] Prochaska JJ, Rossi JS, Redding CA, Rosen AB, Tsoh JY, Humfleet GL, Eisendrath SJ, Meisner MR, Hall SM. Depressed smokers and stage of change: implications for treatment interventions. Drug Alcohol Depend. 2004 Nov 11;76(2):143-51. doi: 10.1016/j.drugalcdep.2004.04.017. PMID 15488338
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Background] Jarvis MJ, Tunstall-Pedoe H, Feyerabend C, Vesey C, Saloojee Y. Comparison of tests used to distinguish smokers from nonsmokers. Am J Public Health. 1987 Nov;77(11):1435-8. doi: 10.2105/ajph.77.11.1435. PMID 3661797
- [Background] Patten CA, Martin JE, Filter KJ, Wolter TD. Utility and accuracy of collateral reports of smoking status among 256 abstinent alcoholic smokers treated for smoking cessation. Addict Behav. 2002 Sep-Oct;27(5):687-96. doi: 10.1016/s0306-4603(01)00202-7. PMID 12201377
- [Background] Adler NE, Epel ES, Castellazzo G, Ickovics JR. Relationship of subjective and objective social status with psychological and physiological functioning: preliminary data in healthy white women. Health Psychol. 2000 Nov;19(6):586-92. doi: 10.1037//0278-6133.19.6.586. PMID 11129362
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] DiClemente CC, Prochaska JO, Fairhurst SK, Velicer WF, Velasquez MM, Rossi JS. The process of smoking cessation: an analysis of precontemplation, contemplation, and preparation stages of change. J Consult Clin Psychol. 1991 Apr;59(2):295-304. doi: 10.1037//0022-006x.59.2.295. PMID 2030191
- [Background] Hall SM, Havassy BE, Wasserman DA. Commitment to abstinence and acute stress in relapse to alcohol, opiates, and nicotine. J Consult Clin Psychol. 1990 Apr;58(2):175-81. doi: 10.1037//0022-006x.58.2.175. PMID 2335634